CLINICAL TRIAL: NCT00132054
Title: Phase I Study of Weekly Irinotecan Combined With Amrubicin in Previously Treated Small-Cell Lung Cancer
Brief Title: Amrubicin and Irinotecan in Treating Patients With Recurrent or Relapsed Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Japan Multinational Trial Organization (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: JMTO-LC03-03; CDR0000439464 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2006-12

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — amrubicin; Irinotecan

INTERVENTIONS:
Drug: amrubicin hydrochloride
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as amrubicin and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of amrubicin when given together with irinotecan in treating patients with recurrent or relapsed extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and maximum tolerated dose of amrubicin when combined with irinotecan in patients with recurrent or relapsed extensive stage small cell lung cancer.

Secondary

* Determine the response rate in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the frequency and severity of adverse events in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of amrubicin.

Patients receive amrubicin on day 1 and irinotecan IV on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of up to 6 patients receive escalating doses of amrubicin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 1/3 (or 33%) of patients experience dose-limiting toxicity. An additional 6 patients are treated at the MTD.

PROJECTED ACCRUAL: A total of 6-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer

  * Extensive stage disease
* Recurrent or relapsed disease after 1-2 prior chemotherapy and/or radiotherapy regimens
* No unmanageable massive pleural effusion or pericardial effusion by chest CT scan
* No symptomatic brain metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.5 g/dL

Hepatic

* ALT and AST ≤ 2 times upper limit of normal
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine normal

Cardiovascular

* No uncontrolled hypertension
* No unstable angina
* No congestive heart failure
* No myocardial infarction within the past year
* No ventricular arrhythmia requiring medical intervention
* No other serious cardiovascular disease

Pulmonary

* Arterial oxygen pressure (PaO_2) ≥ 70 torr
* No interstitial pneumonitis or pulmonary fibrosis by chest x-ray

Gastrointestinal

* No serious diarrhea
* No paralytic or obstructive ileus

Other

* Not pregnant or nursing
* No uncontrolled diabetes
* No severe infectious disorder

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior anthracycline or its derivatives at > the upper dose limit (e.g., daunorubicin ≥ 25 mg/kg, doxorubicin ≥ 500 mg/m^2, or epirubicin ≥ 900 mg/m^2)

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-05; Primary Completion 2006-12 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tadashi Mio, MD, Study Chair — Kyoto University Hospital
Locations (7):
- Japan (7):
  - Gunma Cancer Center, Gunma
  - National Hospital Organization - Dohoku National Hospital, Hokkaido
  - Kyoto University Hospital, Kyoto
  - Kitano Hospital, Osaka
  - Osaka Police Hospital, Osaka
  - Osaka Kosei Nenkin Hospital, Osaka
  - National Hospital Organization - Osaka National Hospital, Osaka